CLINICAL TRIAL: NCT05875012
Title: Effect of Action Observation Physical Training on Quality of Upper Limb and Functional Independence in Children With Hemiplegia
Acronym: AOPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Essam Abdelfattah, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Action observation training
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: HCP

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation arm (Active Comparator)
  Interventions: Other: action observation physical training
- traditional physical training (Active Comparator)
  Interventions: Other: Traditional physical therapy training

INTERVENTIONS:
Other: action observation physical training — Action observation training 3 sessions per week for 3 successive months
  Arms: Action observation arm
Other: Traditional physical therapy training — Traditional physical therapy training 3 sessions per week for 3 successive months
  Arms: traditional physical training

SUMMARY:
30 children with a diagnosis of hemiplegic cerebral palsy

DETAILED DESCRIPTION:
children aged 6-9 years were randomized into 2 groups, control group and study group

ELIGIBILITY:
Inclusion Criteria:

* manual ability classification system level II or III, Modified ashwarth scale 1+ or 2

Exclusion Criteria:

* visual or auditory problems ,fixed deformities

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremity skills test | 3 months
  reliable and valid scale,evaluate quality of upper extremity function in four domains dissociated movement,grasp,weight bearing and protective extension

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, DOkki, Egypt

IPD SHARING:
Plan to Share IPD: No